CLINICAL TRIAL: NCT00536146
Title: Trauma, Stress and Persistence of HPA Dysregulation in Alcoholism
Brief Title: The Stress-Hormone System in Alcohol-Dependent Subjects
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999907216; 07-DK-N216
Record Dates: First submitted 2007-09-26; First posted 2007-09-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-01-29

CONDITIONS: Alcoholism
Keywords: Glucocorticoid; Steroids; Dose-Responsive Curve; EC50; Stress Response; Alcoholism
MeSH Terms: conditions — Alcoholism; Fractures, Stress

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study, conducted at the University of Texas Southwestern Medical Center and the Parkland Hospital in Dallas, will examine the stress hormone system of alcohol-dependent people. This system is weakened in alcohol-addicted people. This study will determine how long it is weakened, whether other hormone systems are also weakened and whether changes in the hormone system are associated with previous trauma or stress.

Healthy normal men and men who are alcohol-dependent may be eligible for this study. Candidates must be between 21 and 60 years of age and have at least a 5-year history of active alcohol dependence. They are screened with a medical history, blood and urine tests and questions about alcohol and drug use, psychiatric problems, history of trauma and recent stress.

Participants undergo the following procedures:

Day 1 - Public Speaking Task

At 6:00 PM subjects have an I.V. line (needle attached to a small plastic tube) inserted into a vein in each arm to draw blood samples and give medication. They are then given a light dinner and then lie down and rest. They rinse their mouth out with water and a drop of lemon juice is placed on their tongue. In 30 to 40 seconds they spit into a funnel attached to a collecting tube. A blood sample is collected to measure levels of cortisol (a stress hormone) ACTH (a hormone responsible for the release of cortisol) and neurosteroids (hormones that affect the brain). Subjects then give a 5-minute speech (telling an ending to a story) and solve a math problem in front of a small group of people. They are then asked how they are feeling. Saliva and blood samples are then collected every 10 minutes for the next 60 minutes.

Day 2 - Cosyntropin Study

At 6:30 p.m. subjects have an I.V. line inserted into a vein in each arm. At 7:45 PM and 8:30 PM saliva is collected as described above. Starting at 7:30 PM, blood samples are collected every 10 minutes until 9:00 PM and then every 20 minutes until 10:00 PM. At 8:00 PM cosyntropin (a medicine that stimulates production of cortisol) is given through the I.V. over 1 minute.

Day 3 - oCRH Study

At 6:30 p.m. subjects have an I.V. line inserted into a vein in each arm. At 7:45 PM and 8:30 PM saliva is collected as described above. Starting at 7:30 PM, blood samples are collected every 10 minutes until 9:00 PM and then every 20 minutes until 10:00 PM. At 8:00 PM ovine CRH (a medicine that stimulates production of cortisol) is given through the I.V. over 1 minute.

Participants may be asked to repeat these studies 3 months later.

DETAILED DESCRIPTION:
The hypothalamic-pituitary-adrenal (HPA) axis provides a key biologic link between the brain and the body's behavioral and physiologic responses to stress, recovery, and adaptation. Both mental trauma and chronic alcohol use may produce disturbances in the HPA response to stress. Thus, changes in this system during a period when there is no alcohol intake may impair the body's ability to mount an appropriate response to environmental stressors, heightening the probability of additional alcohol intake. However, the relationship between trauma, stress, and HPA axis disturbances requires further study. In this study, the NIH investigators will attempt to determine if the sensitivity of glucocorticoid gene induction varies with stress. Blood samples will be obtained at The University of Texas Southwestern Medical Center (TSMC) in collaboration with the Veteran's Affairs Medical Center (VA) at Dallas, Texas under a protocol and consent forms approved by TSMC IRB. Only samples collected as described in the TSMC protocol will be studied at NIH.

ELIGIBILITY:
* INCLUSION CRITERIA:

Alcohol-Dependent Subjects:

Male, 21-60 yrs, DSM-IV diagnosis of alcohol dependence, 4-6 weeks abstinence; Alcohol intake of at least 80 grams of absolute alcohol (approximately one six-pack of beer or one-half pint of 100% proof distilled spirits) on a daily basis for at least two weeks prior to the cessation of drinking. Years drinking: at least 5 yr history of active alcohol dependence; Lifetime drug of choice is alcohol; requesting treatment in long-term residential program.

Healthy Controls:

Thirty men age-matched (plus or minus 5 years) with the patients will be studied. Previous studies have typically used the presence or absence of trauma to define trauma groups. However, these studies have focused on specific types of trauma (i.e. childhood, combat) rather than trauma as a cumulative experience. It is unlikely that we will be able to find subjects who have never experienced any trauma, including the death of loved ones, parental separation, natural disaster, crime, etc. Therefore, we will initially recruit controls without regard to trauma level. Following the recruitment of the first ten subjects, trauma scores will be reviewed. If our control group endorses low levels of trauma, we will direct further recruitment towards a group with at least one self-report of significant lifetime trauma such that at 50 percent of the control population has a least one significant lifetime traumatic event.

Only English-speaking subjects will be included. Several of the study questionnaires are only available in English. In addition, these studies are exploratory and require the induction of anxiety. The investigators at TSMC believe it prudent to assure that all subjects are able to communicate easily with all staff during the fMRI and stress induction. Subjects will be recruited from subjects requesting treatment for alcohol dependence at the Dallas VA but no subjects will be seen at NIH.

EXCLUSION CRITERIA:

Alcohol-Dependent Subjects:

* Primary psychoactive dependence disorder other than alcohol, except nicotine and caffeine.
* Active diagnosis of Axis I Schizophrenia, Mood, or Anxiety Disorders (except PTSD).
* Use of medications known to significantly affect HPA axis functioning or neural activity, including all psychotropics with the previous two weeks (or four weeks for fluoxetine).
* Use of medications known to significantly affect HPA axis functioning or neural activity, including all psychotropics with the previous two weeks (or four weeks for fluoxetine). Patients concomitantly using anxiolytics, antidepressants, opioids, lithium, anticonvulsants, sedative/hypnotics, buspirone, beta blockers, alpha adrenergic drugs, steroids, beta agonists, clonidine, dopamine agonists, naltrexone, acamprosate, or disulfiram will be excluded from the study.
* Any medical conditions that might affect HPA axis functioning or possibly endanger the patient's health or behavioral stability. Medical conditions that might limit cooperation (e.g. dementia) or put the patient at medical risk (i.e. significant hematologic, hepatic, renal, or cardiovascular pathology) will be excluded. Patients with past or present neurologic disorders (i.e. head trauma with loss of consciousness requiring hospitalization, transient ischemic attacks, stroke, tumor, etc.) will be excluded.

Healthy Controls:

* Lifetime history of DSM IV Substance Use Disorder (except Nicotine or Caffeine Dependence) or other Axis I disorder.
* One first-degree family member with a substance use disorder (other than nicotine).
* Medical, psychiatric, and medication exclusions will be the same as those described for the alcohol dependent patients.

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70
Dates: Start 2007-09-24; Study Completion 2009-01-29

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Veterans Affairs Medical Center at Dallas, Dallas, Texas